CLINICAL TRIAL: NCT03621241
Title: Immunophenotyping of Blood Cells in the Diagnosis Work-up of Myelodysplastic Syndromes
Acronym: MODIFY
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2018_843_0010
Record Dates: First submitted 2018-06-07; First posted 2018-08-08 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Flow cytometry — Flow cytometry

SUMMARY:
Myelodysplastic syndromes (MDS) are a heterogeneous group of hematological malignancies characterized by cytopenia(s), dysplasia in one or more major myeloid cell lines and progression to acute leukemia. Morphological analysis of peripheral blood (PB) and bone marrow (BM) remains the cornerstone of the diagnosis. Preliminary studies identified Flow Cytometry (FC) markers on red cells, platelets and circulating leukocytes that are expressed differently in MDS and in controls. However, these markers have been evaluated separately. The investigators propose to test in a large cohort of patients these markers, and to combine the most relevant ones in order to define a PB FC-based diagnosis score that would discriminate between MDS and non-clonal hematopoiesis and would avoid useless bone marrow samples in elderly

ELIGIBILITY:
Inclusion Criteria:

1. Patient who have been orally informed, and given a short written information notice about the study
2. Adult patient>18 years
3. For whom a blood sample analysis is routinely prescribed
4. Presenting cytopenia on at least one lineage according to the 2016 WHO classification (Hemoglobin level<100 g/L and/or platelets <150 G/L and/or Neutrophils<1G/L).
5. For whom a bone marrow analysis for morphology assessment and cytogenetics have to be performed, because of suspicion of MDS.t The results of this bone marrow evaluation will classify the patients in Group 1 (MDS diagnosis) and Group 2 (no MDS according to the 2016 WHO criteria), defining the two populations of this validation cohort for whom the FC score will be calculated.

Exclusion Criteria:

1. Transfused patients (less than 3 months) in RBC or platelets units

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MDS
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
identification of the most relevant combination of FC markers | 0 days
  The main objective is to identify the most relevant combination of FC markers to discriminate between already diagnosed MDS patients and non-MDS patients.

SECONDARY OUTCOMES:
prospective validation of a diagnostic score using pre-identified markers | 0 days
  The secondary objective is to build prospectively a diagnostic score using markers identified

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU Amiens-Picardie, Amiens
  - CHRU Lille, Lille
  - CHU Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No